CLINICAL TRIAL: NCT00307216
Title: Randomized Controlled Trial of the Graduated Recovery Intervention Program for First-Episode Psychosis
Brief Title: Graduated Recovery Intervention Program for Enhancing Treatment for First-Episode Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Penn, PhD, Professor of Psychology, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH071252 (NIH); R34MH071252 (NIH); DATR A2-AISZ
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Psychotic Disorders; Schizophrenia
Keywords: First Episode Psychosis; Early Psychosis; Psychosocial Intervention
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive Graduated Recovery Intervention Program plus treatment as usual
  Interventions: Behavioral: Graduated Recovery Intervention Program (GRIP); Behavioral: Treatment as usual (TAU)
- 2 (Active Comparator): Participants will receive treatment as usual
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Graduated Recovery Intervention Program (GRIP) — GRIP is a manual-based comprehensive psychosocial intervention for people recovering from an initial episode of nonaffective psychosis. The purpose of GRIP is to improve occupational functioning after first-episode psychosis and promote goal pursuit and effective illness self-management. Participants assigned to receive TAU plus GRIP will attend therapy sessions weekly for up to 36 weeks, in addition to routine appointments. GRIP includes four phases, each of which focuses on one of the following topics: engagement and wellness management, substance use, persistent symptoms, and functional recovery.
  Arms: 1
Behavioral: Treatment as usual (TAU) — Participants receiving TAU will meet with their case-manager and health care providers on an as-needed basis.

SUMMARY:
This study will determine the effectiveness of the Graduated Recovery Intervention Program, a manual-based individual therapy program, in enhancing the clinical benefit of routine treatment for individuals recovering from their first episodes of psychosis.

DETAILED DESCRIPTION:
Several mental disorders can be classified as psychotic disorders, such as schizophrenia and manic depression. Psychosis is a defining feature of psychotic disorders, and is characterized by delusions and hallucinations that result in extreme impairment of a person's ability to think clearly. First-episode psychosis refers to the first time someone experiences psychotic symptoms or a psychotic episode. The symptoms can be disturbing and unfamiliar to those who have not previously experienced them. The person experiencing first-episode psychosis may not understand what is happening, and may become confused and distressed. Psychosis is treatable, however, and most people recover. Standard treatment for psychosis entails a combination of behavioral therapy and drug therapy. GRIP is a comprehensive psychosocial intervention for people recovering from an initial episode of non-affective psychosis. The purpose of GRIP is to improve occupational functioning after first-episode psychosis and promote goal pursuit and effective illness self-management. This study will determine the effectiveness of GRIP in enhancing the clinical benefit of routine treatment for individuals recovering from their first episodes of psychosis.

Participants in this study will be randomly assigned to receive either treatment as usual (TAU) or TAU plus GRIP. Participants receiving TAU will meet with their case-manager and health care providers on an as-needed basis. Participants assigned to receive TAU plus GRIP will attend therapy sessions weekly for up to 36 weeks, in addition to routine appointments. GRIP includes four phases, each of which focuses on one of the following topics: engagement and wellness management; substance use; persistent symptoms; and functional recovery. Assessments of social functioning, psychotic symptoms, attitudes toward treatment, substance use, and hospital readmission rate will be assessed at baseline, mid-treatment, post-treatment, and at the follow-up visit 3 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for schizophrenia, schizophreniform disorder, or schizoaffective disorder
* Has been in treatment for psychosis for less than 3 years
* Clinically stable (based on clinician judgement)
* IQ score greater than 70
* Currently receiving keyworker services at UNC Hospital's OASIS program

Exclusion Criteria:

* Organic brain disorder
* Substance-induced psychotic disorder
* Mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Role Functioning Scale | Measured at baseline, post-test, and Month 3 follow-up
Heinrichs-Carpenter Quality of Life Scale (QLS) | Measured at baseline, post-test, and Month 3 follow-up
Multidimensional Scale of Perceived Social Support (MSPSS) | Measured at baseline, post-test, and Month 3 follow-up
Global Functioning Scale | Measured at baseline, post-test, and Month 3 follow-up

SECONDARY OUTCOMES:
Brief Evaluation of Medication Influences and Beliefs | Measured at baseline, post-test, and Month 3 follow-up
Positive and Negative Syndrome Scale (PANSS) | Measured at baseline, post-test, and Month 3 follow-up
Calgary Depression Scale for Schizophrenia (CDSS) | Measured at baseline, post-test, and Month 3 follow-up
Brief Trauma Questionnaire (BTQ) | Measured at baseline, post-test, and Month 3 follow-up
PTSD Checklist (PCL) | Measured at baseline, post-test, and Month 3 follow-up
Alcohol Use Scale and Drug Use Scale (AUS/DUS) | Measured at baseline, post-test, and Month 3 follow-up
Number of hospital admissions | Measured at baseline, post-test, and Month 3 follow-up
Ambiguous Intentions Hostility Questionnaire (AIHQ) | Measured at baseline, post-test, and Month 3 follow-up
Goal attainment ratings | Measured at post-test
Scales of Wellbeing | Measured at baseline, post-test, and Month 3 follow-up
Social Skills Performance Assessment (SSPA) | Measured at baseline, post-test, and Month 3 follow-up
Treatment Compliance Scale (TCS) | Measured at post-test

CONTACTS AND LOCATIONS:
Overall Officials: David L. Penn, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Diana O. Perkins, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals OASIS Program for Early Psychosis, Chapel Hill, North Carolina, United States